CLINICAL TRIAL: NCT03782090
Title: Comparisons of Novel Double-lumen Endobronchial Tube for Blind Lung Isolation Technique With Conventional Double-lumen Endobronchial Tube in Patients Undergoing One-lung Ventilation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 4-2018-0698
Record Dates: First submitted 2018-12-18; First posted 2018-12-20 (Actual); Last update posted 2019-05-20 (Actual); Status verified 2019-05

CONDITIONS: Intubation Tube(Intubation Using Double Lumen Endobronchial Tube)

STUDY DESIGN:
Intervention Model Description: Patients were randomly allocated into either control group (n = 95) or experimental group (n = 95) by a computerized randomization table. In control group, endobronchial intubation is performed using conventional technique with left-sided double-lumen endotracheal tube (Shiley®, Covidien, Mansfield, MA, USA). In experimental group, patients are intubated with novel double-lumen endotracheal tube (Ankor®,Insung Medical, Wonjou, S. Korea).
Who Masked: Participant
Masking Description: Patients, investigators who evaluate complication of intubation are blinded to the study group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Endobronchial intubation using conventional technique with left-sided double-lumen endotracheal tube (Shiley®, Covidien, Mansfield, MA, USA)
  Interventions: Device: Endobronchial intubation
- Experimental (Experimental): Endobronchial intubation using novel left-sided double-lumen endobronchial tube (Ankor®,Insung Medical, Wonjou, S. Korea)
  Interventions: Device: Endobronchial intubation

INTERVENTIONS:
Device: Endobronchial intubation — 1. In control group, endobronchial intubation is performed using conventional technique with left-sided double-lumen endobronchial tube(Shiley®). The tube is introduced into the glottis via direct laryngoscopy. After the tube tip passes the vocal cord, the tube is rotated 90º toward the left. The tube is advanced according to the depth(cm) of the tube calculated by the height of patient(12.5+0.1*height). Afterwards, the depth of the tube is adjusted by the compliance of both lung.
  2. In experimental group, patients are intubated with novel double-lumen endobronchial tube(Ankor®). The tube is introduced into the glottis via direct laryngoscopy. After the tube tip passes the vocal cord, the tube is rotated 90º toward the left. Once the carinal cuff of the tube is passed through the vocal cord of patients, the carinal cuff is inflated with 5-8ml of air. The tube is advanced until the tube stops itself at some point along the tracheobronchial tree. And then the carinal cuff is deflated.

SUMMARY:
The study is prospectively conducted on 190 patients aged between 20 and 85 years, American Society of Anesthesiologists (ASA) physical status I - III, undergoing one-lung ventilation for thoracic surgery. Patients were randomly allocated into either control group (n = 95) or experimental group (n = 95) by a computerized randomization table. The size of endobronchial tube is decided based on the diameter of left main bronchus measured on the CT finding of patients. After induction of general anesthesia, in patients assigned to control group, endobronchial intubation is performed using conventional technique with left-sided double-lumen endobronchial tube (Shiley®, Covidien, Mansfield, MA, USA). In experimental group, patients are intubated with novel double-lumen endobronchial tube (Ankor®,Insung Medical, Wonjou, S. Korea). During intubation, the carina cuff of Ankor® is inflated after the tube is rotated 90º toward the left. The tube is advanced until slight resistance is felt, then the carina cuff is deflated. In both groups, fiberoptic bronchoscope is performed to evaluate the position of endobronchial tube after intubation. If endobronchial tube is not in optimal position, the depth of tube is corrected to optimal position under guidance of fiberoptic bronchoscope. Airway injury is confirmed using fiberoptic bronchoscope before extubation. The success of endobronchial intubation, position of endobronchial tube, the corrected depth of endobronchial tube, time consumption for endobronchial intubation and complication of intubation such as airway injury, pain, and hoarseness are compared between two groups.

ELIGIBILITY:
Inclusion Criteria:

1. ASA classification 1-3
2. aged between 20 to 85
3. undergoing one lung ventilation using left-sided double-lumen endobronchial tube for thoracic surgery

Exclusion Criteria:

1. Expected difficult intubation (neck extension<35 degrees, mandibular-hyoid distance < 6 cm, sternomental distance < 12.5 cm)
2. anomaly of tracheobronchial tree
3. intraluminal lesion in left or right bronchus
4. Obesity (Body Mass Index > 30)
5. upper respiratory infection
6. Thoracic surgical history
7. blood coagulation disorder
8. emergency operation

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2018-09-05 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Optimal position of double-lumen endobronchial tube | 1 day (after intubation)
  On fiberoptic bronchoscopic view after intubation, optimal position of double-lumen endobronchial tube is defined when the bronchial cuff of the tube is immediately below the tracheal carina and there is a clear view of the left subcarina with unobstructed left upper and lower bronchi.

SECONDARY OUTCOMES:
The corrected depth of endobronchial tube | 1 day (after intubation)
  The corrected depth of endobronchial tube is defined as the difference between the depth of endobronchial tube before and after the depth of tube is corrected to optimal position under guidance of fiberoptic.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Severance, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No